CLINICAL TRIAL: NCT01098500
Title: Liver Function Test (LFT) Elevations in Cancer Patients and Users of Tyrosine Kinase Inhibitor (TKI) Drugs Using the LabRx Database
Brief Title: Liver Function Test (LFT) Elevations in Cancer Patients and Users of Tyrosine Kinase Inhibitor (TKI) Drugs
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113153; WEUKSTV3635 (Other: GSK); EPI40661 (Other: GSK)
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: Liver function; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Neoplasms | interventions — Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients: Adults (age ≥18 years) with at least two ICD-9 codes for a particular cancer within a 6 month timeframe and at least one code for a TKI drug that occurs on or after the first cancer diagnosis code
  Interventions: Drug: Tyrosine kinase inhibitors

INTERVENTIONS:
Drug: Tyrosine kinase inhibitors — Lapatinib, erlotinib, gefitinib, dasatinib, imatinib, nilotinib (analyzed as a class of drugs, not by individual drug)

SUMMARY:
A retrospective cohort study using the LabRx medical claims database will be performed to address these objectives. The primary objective of this project is to examine the background rates of liver function test (LFT) abnormalities in cancer patients treated with tyrosine kinase inhibitors (TKIs).

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years) with at least two ICD-9 codes for a particular cancer (ICD-9 code 140-208.9) within a 6 month timeframe and at least one code for a TKI drug that occurs on or after the first cancer diagnosis code
* At least one month (30 days) of enrolment prior to index date and three months (91 days) of follow-up post index date; and
* Continuous enrolment in the LabRx database during follow-up.

Exclusion Criteria:

* Less than 18 years old
* Less than one month (30 days) of enrolment prior to index date or three months (91 days) of follow-up post index date; and
* Not continuously enrolled in the LabRx database during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort study using the LabRx medical claims EMR database. This database contains medical claims information including diagnoses, treatments, medications, and laboratory results for 23.3 million US residents. The study cohort included adult patients (age ≥18 years) with any cancer diagnosed between October 1, 2004-June 1, 2009 who were treated with 1 one or more of the TKI agents-erlotinib, gefitinib, dasatinib, imatinib, nilotinib, or lapatinib. The index date for this cohort was the date of first administration or prescription of the TKI agent on or following the date of the first cancer diagnosis.
Sampling Method: Probability Sample
Enrollment: 3800 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This observational study was conducted and supported by GlaxoSmithKline.
Groups:
- TKI Cohort: Adult (age >=18 years) members of the LabRx database (A United States healthcare claims database containing the aggregated health claims experience of the covered lives managed by United Healthcare) with at least two International Classification of Disease (ICD)-9 codes for any cancer within a six-month timeframe and at least one code for an Epidermal Growth Factor Receptor (EGFR) targeted small molecule tyrosine kinase inhibitor (TKI) drug (erlotinib, gefitinib, dasatinib, imatinib, nilotinib, and lapatinib). TKI initiation must have occurred within 30 days prior to or any time after the first cancer diagnosis. The index date was the date of the first TKI prescription, and patients were followed from 30 days prior to the index date through the last visit in the database (which may be due to death or change in health plan), or the study cut-off date of June 1, 2009, whichever came first.
Period: Overall Study
Arm/Group | TKI Cohort
Started | 3800
Completed | 3800
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TKI Cohort
Number analyzed (Participants) | 3800
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (12)
Sex/Gender, Customized [Number; unit: participants]
  Female | 2061
  Male | 1737
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With ALT (Alanine Transaminase) >=3x (Times) Upper Limit of Normal (ULN)
Description: Prevalence of patients with an ALT elevation >=3x ULN among patients who had liver function testing during the baseline period (30 days prior to initiation of TKI drug).
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had liver function testing within 30 days prior to the initiation of TKI drug.
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 498
participants | 11
Statistical Analysis 1: Comparison: TKI Cohort; Test type: Superiority or Other; Prevalence percentage = 2.2, 95% CI 2-sided [0.9 to 3.5] — Prevalence percentage is the number of patients with an ALT >=3 times ULN divided by all patients that were tested at baseline (30 days prior to initiation of TKI drug)

2. Primary Outcome: Incidence of ALT >=3x ULN
Description: Number of patients with ALT >=3 times ULN among patients with a normal ALT measurement during the baseline period (30 days prior to initiation of TKI drug). Normal is defined as an ALT <1 times ULN at baseline.
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had normal ALT (<1x ULN) during baseline (within 30 days prior to the initiation of TKI drug)
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 344
participants | 18
Statistical Analysis 1: Comparison: TKI Cohort; Test type: Superiority or Other; Incidence Rate (IR) = 6.2, 95% CI 2-sided [3.3 to 9.0] — Incidence rate (IR) is the number of patients with an ALT >=3 times ULN after initiation of TKI divided by person time contributed by all patients with normal ALT (<1 times ULN) at baseline. IR expressed per 100 person years

3. Primary Outcome: Number of Hy's Law Patients (ALT or AST >= 3x ULN and ALP <2x ULN and BIL >= 2x ULN)
Description: Prevalence of patients with Hy's Law (ALT or AST >=3x ULN and ALP <2x ULN and BIL >=2x ULN, where AST = aspartate transaminase, ALP = alkaline phosphatase, BIL= bilirubin) among patients who had liver function testing during the baseline period (30 days prior to initiation of TKI drug).
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had liver function testing within 30 days prior to the initiation of TKI drug).
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 500
participants | 2
Statistical Analysis 1: Comparison: TKI Cohort; Test type: Superiority or Other; Prevalence percentage = 0.4, 95% CI 2-sided [0.1 to 1.4] — Prevalence percentage is the number of patients with Hy's Law divided by all patients that were tested at baseline (30 days prior to initiation of TKI drug)

4. Primary Outcome: Incidence of Hy's Law (ALT or AST >=3x ULN and ALP <2x ULN and BIL >=2x ULN)
Description: Number of patients with Hy's Law (ALT or AST >= 3x ULN and ALP <2x ULN and BIL >= 2x ULN) among patients with normal ALT, AST, ALP, and BIL measurements during the baseline period (30 days prior to initiation of TKI drug). Normal is defined as an ALT AST, ALP, and BIL <1 times ULN at baseline.
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had normal ALT, AST, ALP, and BIL (<1x ULN) during baseline (within 30 days prior to the initiation of TKI drug).
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 307
participants | 1
Statistical Analysis 1: Comparison: TKI Cohort; Test type: Superiority or Other; Incidence Rate (IR) = 0.4, 95% CI 2-sided [0.0 to 2.0] — Incidence rate (IR) is the number of patients with Hy's Law after initiation of TKI divided by person time contributed by all patients with normal ALT, AST, ALP, and BIL (< 1 times ULN) at baseline. IR is expressed per 100 person years

5. Secondary Outcome: Maximum ALT Elevation Reached During Follow-up
Description: Number of patients whose maximum ALT elevation fell within the indicated ULN range among patients with at least one incident ALT elevation during follow-up
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident ALT elevation during follow-up.
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 101
participants
  ALT: >=1x ULN to <3x ULN | 82
  ALT: >=3x ULN to <5x ULN | 8
  ALT: >=5x ULN to <10x ULN | 10
  ALT: >=10x ULN to <20x ULN | 0
  ALT: >=20x ULN | 1

6. Secondary Outcome: Median Time to the Maximum ALT Elevation During Follow-up
Description: Median time (in months) between index date and the date of maximum ALT elevation.
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident ALT elevation during follow-up.
Measure: Median (Full Range); unit: months
Arm/Group | TKI Cohort
Number analyzed (Participants) | 101
months
  ALT: >=1x ULN to <3x ULN | 4 [1 to 42]
  ALT: >=3x ULN to <5x ULN | 8 [0 to 17]
  ALT: >=5x ULN to <10x ULN | 3 [1 to 18]
  ALT: >=10x ULN to <20x | 0 [0 to 0]
  ALT: >=20x ULN | 7 [7 to 7]

7. Secondary Outcome: Maximum AST Elevation Reached During Follow-up
Description: Number of patients whose maximum AST elevation fell within the indicated ULN range among patients with at least one incident AST elevation during follow-up
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident AST elevation during follow-up.
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 101
participants
  AST: >=1x ULN to <3x ULN | 87
  AST: >=3x ULN to <5x ULN | 8
  AST: >=5x ULN to <10x ULN | 3
  AST: >=10x ULN to <20x ULN | 2
  AST: >=20x ULN | 1

8. Secondary Outcome: Median Time to the Maximum AST Elevation During Follow-up
Description: Median time (in months) between index date and date of maximum AST elevation
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident AST elevation during follow-up.
Measure: Median (Full Range); unit: months
Arm/Group | TKI Cohort
Number analyzed (Participants) | 101
months
  AST: >=1x ULN to <3x ULN | 4 [0 to 50]
  AST: >=3x ULN to <5x ULN | 5 [1 to 18]
  AST: >=5x ULN to <10x ULN | 3 [1 to 17]
  AST: >=10x ULN to <20x ULN | 7 [3 to 11]
  AST: >=20x ULN | 7 [7 to 7]

9. Secondary Outcome: Maximum ALP Elevation Reached During Follow-up
Description: Number of patients whose maximum ALP elevation fell within the indicated ULN range among patients with at least one incident ALP elevation during follow-up
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident ALP elevation during follow-up.
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 75
participants
  ALP: >=1x ULN to <2x ULN | 61
  ALP: >=2x ULN to <3x ULN | 7
  ALP: >=3x ULN to <5x ULN | 4
  ALP: >=5x ULN to <10x ULN | 3
  ALP: >=10x ULN | 0

10. Secondary Outcome: Median Time to the Maximum ALP Elevation During Follow-up
Description: Median time (in months) between index date and date of maximum ALP elevation
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident ALP elevation during follow-up.
Measure: Median (Full Range); unit: months
Arm/Group | TKI Cohort
Number analyzed (Participants) | 75
months
  ALP: >=1x ULN to <2x ULN | 5 [0 to 34]
  ALP: >=2x ULN to <3x ULN | 3 [0 to 5]
  ALP: >=3x ULN to <5x ULN | 11 [3 to 17]
  ALP: >=5x ULN to <10x ULN | 8 [3 to 11]
  ALP: >=10x ULN | 0 [0 to 0]

11. Secondary Outcome: Maximum BIL Elevation Reached During Follow-up
Description: Number of patients whose maximum BIL elevations fell within the indicated ULN range among patients with at least one incident BIL elevation during follow-up
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident BIL elevation during follow-up.
Measure: Number; unit: participants
Arm/Group | TKI Cohort
Number analyzed (Participants) | 70
participants
  BIL: >=1x ULN to <1.5x ULN | 46
  BIL: >=1.5x ULN to <2x ULN | 9
  BIL: >=2x ULN to <5x ULN | 8
  BIL: >=5x ULN to <10x ULN | 4
  BIL: >=10x ULN | 3

12. Secondary Outcome: Median Time to the Maximum BIL Elevation During Follow-up
Description: Median time (in months) between index date and date of maximum BIL elevation
Time Frame: Study period was October 1, 2004-June 30, 2009. Patients had at least 91 days of follow-up post index date.
Population: Members of the TKI cohort who had at least one incident BIL elevation during follow-up.
Measure: Median (Full Range); unit: months
Arm/Group | TKI Cohort
Number analyzed (Participants) | 70
months
  BIL: >=1x ULN to <1.5x ULN | 3 [0 to 26]
  BIL: >=1.5x ULN to <2x ULN | 3 [0 to 33]
  BIL: >=2x ULN to <5x ULN | 4 [2 to 17]
  BIL: >=5x ULN to <10x ULN | 8 [5 to 11]
  BIL: >=10x ULN | 6 [2 to 18]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | TKI Cohort
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.